CLINICAL TRIAL: NCT03911986
Title: Risk-Based Screening for the Evaluation of Atrial Fibrillation Trial (R-BEAT)
Brief Title: Risk-Based Screening for the Evaluation of Atrial Fibrillation Trial
Acronym: R-BEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Ruairi Waters, Associate Specialist in Stroke Medicine, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 17-CRFG 17
Record Dates: First submitted 2018-03-21; First posted 2019-04-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation and Flutter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A randomized controlled cross-over multi-centered clinical trial in General Practice, comparing; a) opportunistic pulse screening + immediate ELR device (R-Test) for 1 week; or, b) opportunistic pulse screening + delayed ELR device (R-Test) for 1 week, in patients with CHA2DS2-VASc score of 3 or greater, and without a contraindication to oral anticoagulation.
Masking Description: There is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate External Loop Recorder (Other): Participants randomized to the Immediate External Loop Recorder group will be monitored for the duration of the first week of the study using the Novacor R-Test 4.
  Interventions: Device: R Test 4 External Loop Recorder
- Delayed External Loop Recorder (Other): Participants randomized to the Delayed External Loop Recorder group will be monitored for the duration of the second week of the study using the Novacor R-Test 4.
  Interventions: Device: R Test 4 External Loop Recorder

INTERVENTIONS:
Device: R Test 4 External Loop Recorder — The R-Test 4 is an externally worn, re-usable, battery-powered, lightweight ECG monitor, which records events triggered by cardiac arrhythmias. It is worn for 7 days. Cardiac monitoring is triggered by tachycardia or detection of irregular pulses or patient may trigger recording, if the participant experience symptoms (e.g. palpitations). The patient wears 2 chest leads (on one, the R-Test device is attached, weight 42g). The R-Test 4 is CE marked, and uses an FDA-approved algorithm for automatic detection of atrial fibrillation, and permits 5 minutes of pre-event recording and 5 minutes of post-event recording.

SUMMARY:
1. To determine whether a risk-based screening programme for occult paroxysmal atrial fibrillation, involving extended cardiac monitoring in adults with CHA2DS2-VASc score of 3 or greater, increases the detection of new atrial fibrillation/flutter.
2. To determine whether a risk-based screening programme for occult paroxysmal atrial fibrillation, involving extended cardiac monitoring in adults with CHA2DS2-VASc score of 3 or greater, is cost-effective.
3. To determine the sensitivity, specificity, positive predictive value and negative predictive values of self-monitoring of pulse in adults for detection of atrial fibrillation.
4. To determine the cost, cost effectiveness, and budget impact of a risk-based screening programme for occult paroxysmal atrial fibrillation, relative to a control of usual care in general practice.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability. A first diagnosis of atrial fibrillation may occur at the time of stroke (e.g. about 45% of patients with acute stroke). Undiagnosed atrial fibrillation is therefore a major care-gap in stroke prevention.

Against this backdrop, oral anticoagulant therapy is extremely effective at reducing the risk of ischemic stroke in atrial fibrillation, associated with a two-thirds risk reduction. Therefore, a major care gap in stroke prevention is the prevalence of undetected atrial fibrillation in the community. Traditional pulse screening in all patients > 65 years detects new atrial fibrillation in about 1% of people.

The CHA2DS2-VASc score was developed and validated to risk-stratify patients with atrial fibrillation into low, intermediate and high risk of stroke. The Investigators believe that the CHA2DS2-VASc score represents an opportunity to identify patients at high risk of atrial fibrillation, but also identifies this at highest risk of stroke, and therefore those that will derive greatest benefit from anticoagulant therapy.

The advent of external-worn event loop recorders (ELRs) present a more convenient and efficient method of detecting atrial fibrillation. Loop recorders have an in-built diagnostic algorithm that identifies atrial fibrillation, and initiates recordings before and after the event-trigger. This rhythm strip is then examined and confirmed by the trial cardiac technician. The investigators will examine if using external loop recorders in patients identified as high risk will improve the detection rate of paroxysmal atrial fibrillation.

The study is a randomised controlled cross-over multi-centered clinical trial in General Practice. Ethical approval has been sought from the Galway University Hospitals research ethics committee. The investigators have also engaged with Clinical Research Patient and Public Involvement.

The investigators primary research question is whether extended cardiac rhythm monitoring (with ELR for 1 week), compared to standard care, in patients pre-identified to be at high-risk of atrial fibrillation (defined by CHA2DS2-VASc score >2) increases the detection of new atrial fibrillation resulting in introduction of oral anticoagulant therapy, that is efficient, acceptable to patients and cost-effective.

All participating general practices will require the Socrates software package. The investigators will run analyses to identify patients with a CHA2DS2-VASc of 3 or greater. The investigators will exclude all patients with known atrial fibrillation, those in whom contraindications to oral anticoagulant therapy exist, and those who are deemed unsuitable for extended monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a study specific Informed Consent Form
2. 55 years of age or older
3. Attending one of the participating General Practices in the R-BEAT Trial
4. Attended at least one GP appointment within the past 12 months
5. CHA2DS2-VASc Score >2

Exclusion Criteria:

1. Contraindication to oral anticoagulant therapy

   1. History of intracerebral haemorrhage
   2. Prior intolerance or refusal of oral anticoagulant therapy

      *(If intolerant or refused warfarin, may be included if considered suitable for non vitamin-K oral anticoagulant, NOAC)
   3. Gastrointestinal haemorrhage of unexplained or unmodifiable aetiology (i.e. risk of haemorrhage has not been reduced)
   4. Other major bleed that would exclude oral anticoagulant therapy
2. Known Atrial fibrillation/flutter
3. Currently prescribed oral anticoagulant therapy
4. Unsuitable for anticoagulant therapy, in opinion of attending general practitioner
5. Unsuitable for cardiac monitoring, in opinion of attending general practitioner
6. Allergies to plasters or adhesives
7. Has had cardiac monitoring for >48 hours within the last 12 months, has an implantable loop recorder, or scheduled to have cardiac monitoring/ILR.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
New detected (and centrally confirmed) cases of atrial fibrillation/flutter > 2 minutes | 2 years
  New detected (and centrally confirmed) cases of atrial fibrillation/flutter > 2 minutes in duration using a built in diagnostic algorithm that identifies probable atrial fibrillation. The identified instances will be reviewed by a cardiologist for confirmation of atrial fibrillation/atrial flutter

SECONDARY OUTCOMES:
Initiation of oral anticoagulation | 3 months
  prescription

CONTACTS AND LOCATIONS:
Overall Officials: Colin Hardy, BSc, Study Chair — Project Officer and Site Management Coordinator
Locations (1):
- HRB Clinical Research Facility Galway, Galway, County Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy R, Waters R, Murphy A, McDermott S, Reddin C, Hernon O, Davies N, Alvarez-Iglesias A, Twomey E, O'Shea E, Sloane P, Curran J, Kiely A, Waters C, Kilraine J, McDonagh S, Carney A, Devane D, O'Donnell M. Risk-based screening for the evaluation of atrial fibrillation in general practice (R-BEAT): a randomized cross-over trial. QJM. 2025 Mar 1;118(3):166-173. doi: 10.1093/qjmed/hcaf001. PMID 39786890